CLINICAL TRIAL: NCT02220907
Title: Long-term Administration Study of MT-2412 in Patients With Type 2 Diabetes Mellitus
Brief Title: Long-Term Safety Study of MT-2412 in Japanese Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-2412-J01
Record Dates: First submitted 2014-08-19; First posted 2014-08-20 (Estimated); Results first posted 2018-08-16 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: MT-2412; MP-513; TA-7284; Teneligliptin; Canagliflozin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-(4-(4-(3-methyl-1-phenyl-1H-pyrazol-5-yl)piperazin-1-yl)pyrrolidin-2-ylcarbonyl)thiazolidine; Canagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Teneligliptin/Canagliflozin (Experimental): Patients receive Teneligliptin and Canagliflozin once daily for 52 weeks.
  Interventions: Drug: Teneligliptin/Canagliflozin

INTERVENTIONS:
Drug: Teneligliptin/Canagliflozin — Co-administration of Teneligliptin and Canagliflozin orally once daily for 52 weeks.
  Other Names: Tenelia; MP-513; Canaglu; TA-7284

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of co-administration of Teneligliptin (MP-513) and Canagliflozin (TA-7284) once daily for 52 weeks in Japanese patients with Type 2 diabetes mellitus who are receiving treatment with Teneligliptin and have inadequate glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Men or women age ≥20 years old
* HbA1c of ≥7.0% and <10.5%
* FPG of ≤ 270 mg/dL
* Patients who are under dietary management and taking therapeutic exercise for diabetes over 12 weeks before treatment period

Exclusion Criteria:

* Patients with type I diabetes, diabetes mellitus resulting from pancreatic disorder, or secondary diabetes
* Patients with serious diabetic complications
* Patients with hereditary glucose-galactose malabsorption or primary renal glucosuria
* Patients with Class III/IV heart failure symptoms according to New York Heart Association (NYHA) functional classification
* Patients with severe hepatic disorder or severe renal disorder.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2014-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Kadowaki, MD, Study Director — Tokyo University; Nobuya Inagaki, MD, Study Director — Kyoto University; Kazuoki Kondo, MD, Study Director — Tanabe Pharma Corporation
Locations (6):
- Japan (6):
  - Research site, Chugoku
  - Research site, Chūbu
  - Research site, Hokkaido
  - Research site, Kanto
  - Research site, Kyushu
  - Research site, Tōhoku

REFERENCES:
- [Result] Kadowaki T, Inagaki N, Kondo K, Nishimura K, Kaneko G, Maruyama N, Nakanishi N, Watanabe Y, Gouda M, Iijima H. Long-term safety and efficacy of canagliflozin as add-on therapy to teneligliptin in Japanese patients with type 2 diabetes. Diabetes Obes Metab. 2018 Jan;20(1):77-84. doi: 10.1111/dom.13038. Epub 2017 Jul 31. PMID 28608617

RESULTS

PARTICIPANT FLOW:
Groups:
- Teneligliptin+Canagliflozin: Teneligliptin and Canagliflozin once daily for 52 weeks.
Period: Overall Study
Arm/Group | Teneligliptin+Canagliflozin
Started | 153
Completed | 142
Not Completed | 11
Not completed — Adverse Event | 7
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2
Not completed — Conflict with the stopping criteria | 1

BASELINE CHARACTERISTICS:
Arm/Group | Teneligliptin+Canagliflozin
Number analyzed (Participants) | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 119
  >=65 years | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 108

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: 52 Weeks
Measure: Number; unit: participants
Arm/Group | Teneligliptin+Canagliflozin
Number analyzed (Participants) | 153
participants
  Serious Adverse Event | 11
  Adverse Event | 107

2. Secondary Outcome: Change From Baseline in Percentage of Glycated Hemoglobin (HbA1c)
Description: The change from baseline in percentage of HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Week 52.
Time Frame: Baseline, 52 Weeks
Population: Full analysis set, last observation carried forward
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Teneligliptin+Canagliflozin
Number analyzed (Participants) | 153
percentage of HbA1c | -0.99 (0.84)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose Level
Description: The change from baseline in fasting plasma glucose level collected at Week 52.
Time Frame: Baseline, 52 Weeks
Population: Full analysis set, last observation carried forward. Outcome measure for one patient was not assessed at a certain timepoint due to dropout.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Teneligliptin+Canagliflozin
Number analyzed (Participants) | 152
mg/dL | -38.6 (29.8)

4. Secondary Outcome: Percentage Change in Body Weight From Baseline
Description: The percentage change from baseline in body weight collected at Week 52.
Time Frame: Baseline, 52 Weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Teneligliptin+Canagliflozin
Number analyzed (Participants) | 152
percent change | -3.92 (3.81)

ADVERSE EVENTS:
Arm/Group | Teneligliptin+Canagliflozin
Serious Adverse Events (participants affected / at risk) | 11/153
Other Adverse Events (participants affected / at risk) | 61/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Teneligliptin+Canagliflozin (N=153)
Influenza (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Herpes zoster disseminated (Infections and infestations) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cataract (Eye disorders) | 2
Myocardial infarction (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Sinus node dysfunction (Cardiac disorders) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Teneligliptin+Canagliflozin (N=153)
Nasopharyngitis (Infections and infestations) | 47
Constipation (Gastrointestinal disorders) | 8
Eczema (Skin and subcutaneous tissue disorders) | 8
Pollakiuria (Renal and urinary disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other